CLINICAL TRIAL: NCT04897620
Title: COMPARISON OF SYSTEMIC INFLAMMATION-RELATED HEMATOLOGICAL PARAMETERS IN ACUTE AND CHRONIC LOW BACK PAIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Elzem Bolkan Günaydın, Lecturer Doctor, Ufuk University
Other Study IDs: 2021-06-10
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Scanning the blood test results — Participants' age, gender, duration of low back pain (days), if evaluated, conditions associated with low back pain in cases with subacute/chronic pain, ESR, CRP, RDW, MPV, neutrophil count, lymphocyte count, eosinophil count and platelet count in blood tests at admission examinations were recorded. NLR was calculated by dividing the number of neutrophils by the number of lymphocytes, PLR by dividing the number of platelets by the number of lymphocytes, ELR by dividing the number of eosinophils by the number of lymphocytes, and SII by the formula "platelet numberxneutrophil number/lymphocyte number"

SUMMARY:
The aim of the study is to compare the neutrophils to lymphocytes ratio (NLR), platelets to lymphocytes ratio (PLR), eosinophils to lymphocytes ratio (ELR), red blood cell distribution width (RDW), mean platelet volume (MPV), systemic immune inflammation index (SII), erythrocyte sedimentation rate (ESR) and C reactive protein (CRP) which are the hematological parameters associated with systemic inflammation in acute and subacute/chronic low back pain. Secondary purpose; evaluation of the prognostic roles of hematological parameters associated with systemic inflammation in low back pain in predicting chronicity.This study is a retrospective case-control study. The data of patients who applied to the emergency department with the complaint of acute (less than 4 weeks) low back pain or to the Physical Medicine and Rehabilitation outpatient clinic with the complaint of subacute (lasting 4-12 weeks) or chronic (longer than 12 weeks) non-specific low back pain in the last 3 years will be scanned. The data of patients who applied with complaints other than medical conditions known to be associated with painful conditions and/or inflammatory response will be screened as a control group. The data of patients between the ages of 18-65 will be included in the study. In conclusion, the data of 150 patients who presented with acute non-specific low back pain, 150 patients who presented with subacute/chronic non-specific low back pain and 150 participants as the control group will be included in the study for use in analysis. Participants' age, gender, duration of low back pain (days), if evaluated, conditions associated with low back pain in cases with subacute/chronic pain, ESR, CRP, RDW, MPV, neutrophil count, lymphocyte count, eosinophil count and platelet count in blood tests at admission examinations will be recorded. NLR will be calculated by dividing the number of neutrophils by the number of lymphocytes, PLR by dividing the number of platelets by the number of lymphocytes, ELR by dividing the number of eosinophils by the number of lymphocytes, and SII by the formula "platelet numberxneutrophil number/lymphocyte number".

ELIGIBILITY:
Inclusion Criteria:

* The data of patients who applied to the emergency department with the complaint of acute (less than 4 weeks) low back pain or to the Physical Medicine and Rehabilitation outpatient clinic with the complaint of subacute (lasting 4-12 weeks) or chronic (longer than 12 weeks) non-specific low back pain in the last 3 years.
* The data of patients between the ages of 18-65.

Exclusion Criteria:

* Patients who have systemic diseases or internal organ pathologies that may cause low back pain, acute/chronic infection, malignancy, rheumatic disease or systemic diseases that may change the hematological inflammation parameters, which are evaluation parameters,
* Patients who have severe neurological involvement findings in imaging examinations or clinical examination,
* Patients who have a history of surgical procedures for the lumbar region in the last 6 months
* Patients those missing one or more of the parameters planned to be evaluated within the scope of the screened data.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The data of patients between the ages of 18-65 who applied to the emergency department with the complaint of acute (less than 4 weeks) low back pain or to the Physical Medicine and Rehabilitation outpatient clinic with the complaint of subacute (lasting 4-12 weeks) or chronic (longer than 12 weeks) non-specific low back pain in the last 3 years will be scanned. The data of patients who applied with complaints other than medical conditions known to be associated with painful conditions and/or inflammatory response will be screened as a control group.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-06-05 (Estimated); Study Completion 2021-06-05 (Estimated)

PRIMARY OUTCOMES:
Erythrocyte sedimentation rate | 1 month
  The erythrocyte sedimentation rate value in blood tests at admission examinations.
C reactive protein | 1 month
  The C reactive protein value in blood tests at admission examinations.
Red blood cell distribution width | 1 month
  The red blood cell distribution width value in blood tests at admission examinations.
Mean platelet volume | 1 month
  The mean platelet volume value in blood tests at admission examinations.
Neutrophils to lymphocytes ratio (NLR) | 1 month
  NLR is calculated by dividing the number of neutrophils by the number of lymphocytes.
Platelets to lymphocytes ratio (PLR) | 1 month
  PLR is calculated by dividing the number of platelets by the number of lymphocytes.
Eosinophils to lymphocytes ratio (ELR) | 1 month
  ELR is calculated by dividing the number of eosinophils by the number of lymphocytes.
Systemic immune inflammation index (SII) | 1 month
  SII is calculated by the formula "platelet numberxneutrophil number/lymphocyte number.

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided